CLINICAL TRIAL: NCT01284972
Title: Short to Mid Term Follow-up of Patient Implanted With the HINTEGRA® Total Ankle Prosthesis
Brief Title: HINTEGRA Total Ankle Prosthesis Follow-up
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-02
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Total Ankle Prosthesis

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HINTEGRA: Patient Implanted with the HINTEGRA Total Ankle Prosthesis more than 2 years ago

SUMMARY:
The Hintegra® Total Ankle Prosthesis is a non constrained, three-component prosthesis that consists of a flat tibial component, an anatomically-shaped talar component, and a high-density polyethylene inlay. The Hintegra ankle was specifically developed as an attempt to address the needs of minimal bone resection, extended bone support, proper ligament balancing, and minimal contact stressed within and around the prosthesis.

The objective of this study is to evaluate the safety and efficacy of the HINTEGRA® Total Ankle prosthesis at short and mid term follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with an Hintegra® Total Ankle Prosthesis (only prosthesis designed with pegs) in primary ankle surgery since a minimum of 2 years
* Age ≥ 18 years
* Have willingness to give his/her data transfer authorisation

Exclusion Criteria:

* History of prior mental illness or patient demonstrates that their mental capacity may interfere with their ability to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient implanted with an Hintegra® Total Ankle Prosthesis (only prosthesis designed with pegs) in primary ankle surgery since a minimum of 2 years
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
rate of device related complications at the follow up after 2 years of implantation | more than 2 years after the implantation

SECONDARY OUTCOMES:
AOFAS Ankle-Hindfoot Scale score (American Orthopaedic Foot and Ankle Society). | more than 2 years after the implantation

CONTACTS AND LOCATIONS:
Locations (6):
- Medical University of Innsbruck, Innsbruck, Austria
- St. Michael's Hospital, Toronto, Canada
- CHU d'Amiens - Hopital Nord, Amiens, France
- AukammKlinik, Wiesbaden, Germany
- Severance Hospital - Yonsei University, Seoul, South Korea
- Hopital San Rafael, Barcelona, Spain